CLINICAL TRIAL: NCT05651295
Title: A Precision Medicine Approach to Target Engagement for Emotion Regulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Matthew Southward (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Matthew Southward, Research Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 64865; K23MH126211 (NIH)
Record Dates: First submitted 2022-12-01; First posted 2022-12-15 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Emotional Regulation; Depression; Anxiety; Borderline Personality Disorder; Obsessive-Compulsive Disorder; Posttraumatic Stress Disorder; Eating Disorders
Keywords: cognitive-behavior therapy; mechanism; ecological momentary assessment; personalization
MeSH Terms: conditions — Emotional Regulation; Depression; Anxiety Disorders; Borderline Personality Disorder; Obsessive-Compulsive Disorder; Stress Disorders, Post-Traumatic; Feeding and Eating Disorders | interventions — Cognitive Restructuring; Mindfulness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Condition (Active Comparator): Participants will learn one of three emotion regulation skills (i.e., cognitive restructuring, opposite to emotion action, mindfulness) that is their personal strength, based on pre-Baseline emotion regulation capacities. They will watch an interactive video, created for the current study, in which they are taught the skill that is their personal strength. They will also be asked to complete a survey during the video in which they will input their own examples to practice the skill and to ensure attention to and comprehension of the material.
  Interventions: Behavioral: Checking the Facts; Behavioral: Opposite to Emotion Action; Behavioral: Mindfulness of Current Emotions
- Standardized Condition (Active Comparator): Participants will learn all three ER skills: cognitive restructuring, opposite to emotion action, and mindfulness. Participants will be asked to watch three interactive videos that cover each skill to provide an analogue to clinical practice in which clinicians must choose whether to provide greater breadth or depth of skill coverage. These videos will be presented in a randomized order and will include the same surveys for attention and comprehension used in the Personalized Condition.
  Interventions: Behavioral: Checking the Facts; Behavioral: Opposite to Emotion Action; Behavioral: Mindfulness of Current Emotions

INTERVENTIONS:
Behavioral: Checking the Facts — Checking the Facts is a form of cognitive reappraisal in which participants identify negatively-valenced automatic thoughts and both generate and consider evidence that challenges the validity of those thoughts.
  Other Names: cognitive restructuring
Behavioral: Opposite to Emotion Action — Opposite to Emotion Action teaches participants to identify their momentary emotion(s), identify the associated behavioral urge(s), and implement a behavior inconsistent with that urge (e.g., approaching a feared stimulus instead of avoiding it).
  Other Names: Opposite Action
Behavioral: Mindfulness of Current Emotions — Mindfulness of Current Emotions teaches participants to nonjudgmentally observe the experience of their emotions, including physiological and cognitive responses to those emotions.
  Other Names: mindfulness; acceptance

SUMMARY:
The proposed study is designed to first test whether teaching people personalized or standardized emotion regulation skills leads to greater decreases in daily negative emotion intensity. Second, using data from an initial sample, the investigators will prospectively assign an independent sample of participants to receive their predicted optimal or non-optimal skills to determine if it is feasible and efficacious to match participants to the most appropriate training condition. Results of these studies may identify the mechanisms by which emotion regulation interventions impact emotional functioning and allow for the development of personalized, evidence-based, and scalable emotion regulation interventions.

ELIGIBILITY:
Inclusion Criteria:

* Elevated emotion dysregulation

Exclusion Criteria:

* Lack of proficiency in English
* No access to smartphone
* Conditions requiring greater than outpatient care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Positive and Negative Affect Schedule-Short Form | 7 times per day for 42 days
  A self-report measure designed to assess the intensity of momentary negative affect. Scores range from 1 to 5, with higher scores indicating greater negative affect and lower scores indicating less negative affect.

SECONDARY OUTCOMES:
Changes in Hamilton Depression Rating Scale | Once every 2 weeks for 6 weeks (4 times total)
  A 17-item clinician-rated measure of the severity and frequency of depressive symptoms over the prior week. Scores range from 0 to 51, with higher scores indicating greater severity and frequency of depressive symptoms and lower scores indicating less severe or frequent depressive symptoms.
Changes in Hamilton Anxiety Rating Scale | Once every 2 weeks for 6 weeks (4 times total)
  A 14-item clinician-rated measure of the severity and frequency of anxiety symptoms over the prior week. Scores range from 0 to 56, with higher scores indicating greater severity and frequency of anxiety symptoms and lower scores indicating less severe or frequent anxiety symptoms.
Changes in Five-Factor Model Score Sheet | Once every 2 weeks for 6 weeks (4 times total)
  A 30-item clinician-rated measure of adaptive and maladaptive variants of the Big Five personality dimensions. Each item is rated from 1-7, with higher scores indicating more maladaptive variants of each Big Five personality dimension and lower scores indicating more adaptive variants of each Big Five personality dimension.
Changes in Ways of Responding Scale | Once every 2 weeks for 6 weeks (4 times total)
  Ratings, made by independent coders masked to participant and condition information, of the quality of written responses to 6 hypothetical stressful scenarios. Scores range from 1-7, with higher scores indicating higher quality responses and lower scores indicating lower quality responses.
Changes in Opposite to Emotion Action Task | Once every 2 weeks for 6 weeks (4 times total)
  A behavioral task in which participants are asked to act in ways that are inconsistent with difficult emotions in response to emotion inductions. Before and after each trial, participants will rate the intensity of their negative emotions using the PANAS Basic Negative Emotion scale, which is a self-report measure designed to assess the intensity of momentary negative affect. Scores range from 1 to 5, with higher scores indicating greater negative affect and lower scores indicating less negative affect.
Changes in Breath-Counting Task | Once every 2 weeks for 6 weeks (4 times total)
  A behavioral and psychophysiological task in which participants will use a keyboard to record how frequently they breathe during a 15-minute period, which will be compared to physiological recordings of breathing rates for accuracy. Scores range from 0-100%, with higher scores indicate greater accuracy and lower scores indicating lower accuracy.
Changes in emotion regulation effectiveness | 7 times per day for 48 days
  A one-item rating of the perceived effectiveness of participants' emotion regulation skills since the previous notification. Scores range from 0 to 4, with higher scores indicating greater effectiveness of the regulation and lower scores indicating less effectiveness of the regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Southward, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No